CLINICAL TRIAL: NCT05089812
Title: The Effect of Platelet-rich Fibrin on Clinical and Patient-centered Outcomes of Third Molar Extractions
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK: 33-451 ex 20/21
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Oral Surgery

STUDY DESIGN:
Intervention Model Description: split-mouth study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test-Group (Experimental): PRF-Group
  Interventions: Procedure: Third-molar extraction using platelet-rich fibrin as a filling of the alveolus
- Control-Group (Placebo Comparator)
  Interventions: Procedure: Third-molar extraction using platelet-rich fibrin as a filling of the alveolus

INTERVENTIONS:
Procedure: Third-molar extraction using platelet-rich fibrin as a filling of the alveolus — see above

SUMMARY:
The fear of oral surgeries is mostly dedicated to pain and swelling in the following days. It is not surprising, that it is of high interest to do anything to reduce these consequences. Maybe this is a reason, why using platelet concentrates in oral health rehabilitation has become common in the last couple of years. Less swelling, less pain, quicker healing. The aims of the present study are to determine the effect of a platelet rich fibrin on postsurgical inflammatory complications and patient-centred outcomes and perceptions, in patients undergoing third molar extractions by split mouth technique.

25 medically healthy adults will be assigned to one of 2 groups (1 test- and 1 control group). This means due to the split mouth technique patients undergo a third molar extraction twice. The first time the patient will be randomly assigned to the test- or control group and the second time the patient will be in the other group (test or control group).

The test groups socket will be filled with a PRF (platelet-rich fibrin)-Clot before suturing the wound during third molar surgery. As well, a blood count and coagulations values will be determined. The control group will be operated conventionally. Swelling will be measured at day 1, 3 and 7 post surgery by CBCT (cone-beam computed tomography) facial scan. Subjects will be examined clinically by examiners at the seventh day after surgery for postoperative complications. In addition, Visual analogue scores (VAS) on pain, swelling and bleeding will be obtained from the patients from day 0 through day 7. The present study will answer an important clinical question with regards to the recommendation of platelet-rich fibrin usage to prevent post-operative complications with third molar surgery and to recommend a platelet-rich fibrin, if required.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy adult [ASA (American Society of Anesthesiologists) classification I-II], age ≥ 16 years old
* Preferably non-smoker, or previous smoker (quit ≥ 5 years), light smoker with less than 20 cigarettes/ day
* Therapeutic or strategic indications
* No allergies against local anasthesia (Articain, Mepivacain) and their preservatives (Natriummetabisulfid E223, natriumchlorid)
* Written consent of the patient
* No infected upper and lower third molars
* Third molars in 4 quadrants and located in maxilla/mandible (classification of Pell and Gregory/ Winter) and indication for extractions

Exclusion Criteria:

* Medically compromised subjects (ASA classification III-V)
* General contraindications against third molar extractions (e.g. immunodeficiency, advanced systemic diseases, corticosteroid medication)
* Treatment or diseases that may have an effect on bone turnover or bone or non-mineralized tissue metabolism (e.g. Bisphosphonates or local radio-therapy)
* Patients with anticoagulant therapy
* Heavy smoker or previous heavy smoker (quit < 5 years; ≥ 20 cigarettes/day)
* Use of any form of antibiotics in the last 3 months or subjects requiring antibiotic prophylaxis prior to dental treatment
* Pregnant or breast feeding. Self declared intend to conceive. A pregnancy test performed for female patients.
* Subjects aged < 16 years old

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Swelling | Pre-surgical and at day 1, 3, 7 and 14 post-surgical
  Buccal swelling will be measured manually as well as within creating a 3D face scan pre-surgical and at day 1, 3, 7 and 14 post-surgical. Scans will be superimposed and compared with Romexis software. Manual measurement: Lines between lateral corner of the eye- jaw angle, Tragus- outer Mouth corner, Tragus-Pogonion will be measured in mm and be compared pre-surgical and at day 1, 3, 7 and 14 post-surgical. longer lines suggest more swelling and a worse outcome.

SECONDARY OUTCOMES:
Change in Inflammatory Complications - Amount of clinical recordings | Pre-surgical and at day 1, 3, 7 and 14 post-surgical
  Clinical recordings of post-surgical inflammatory complications (like issue of purulent matter, restriction of the opening of the mouth, clinical attachment loss of second molar distal, flap closure)
Change in Inflammatory Complications - VAS Swelling | Pre-surgical and at day 1, 3, 7 and 14 post-surgical
  VAS-Scale day 1-7 (Swelling). Scale from 0-10 (0 is no swelling/good outcome, 10 is a very high amount of swelling/bad outcome)
Change in Inflammatory Complications - VAS Bleeding | Pre-surgical and at day 1, 3, 7 and 14 post-surgical
  VAS-Scale day 1-7 (Bleeding) (0 is no bleeding/good outcome, 10 is a very high amount of bleeding/bad outcome)
Change in Inflammatory Complications - VAS Pain | Pre-surgical and at day 1, 3, 7 and 14 post-surgical
  VAS-Scale day 1-7 (pain) (0 is no pain/good outcome, 10 is a very bad pain/bad outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styra, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwittnig K, Kirnbauer B, Truschnegg A, Jakse N, Wolf A, Sokolowski A, Mischak I, Payer M. Effectiveness of platelet-rich fibrin in third molar extractions: a randomized controlled split-mouth study. Clin Oral Investig. 2024 Oct 29;28(11):615. doi: 10.1007/s00784-024-06002-9. PMID 39467892